CLINICAL TRIAL: NCT04190160
Title: Unicenter Interventional Study Aimed at Improving the Quality of Life in a Group of Very Old Patients With Type 2 Diabetes With Fixed-ratio Combination of Insulin Degludec and Liraglutide (iDegLira)
Brief Title: Quality of Life and Fixed-ratio Combination of Insulin Degludec and Liraglutide (iDegLira)
Acronym: XETD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stefano Rizza (Other)
Responsible Party: Sponsor-Investigator, Stefano Rizza, Principal Investigator, University of Rome Tor Vergata
Organization: University of Rome Tor Vergata (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 141/18 XETD2
Record Dates: First submitted 2019-12-01; First posted 2019-12-09 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Type2 Diabetes
Keywords: elderly, diabetes, safety, quality of life
MeSH Terms: conditions — Diabetes Mellitus | interventions — IDegLira

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6 months treatment (Experimental): replacement of whatever pre-existing hypoglicaemic therapeutic scheme, with or without insulin, with a single daily and flexible administration of IDegLira in a pilot little group of very old diabetic patients
  Interventions: Drug: IDegLira

INTERVENTIONS:
Drug: IDegLira — A single administration of IDegLira, dose depending on glicaemic control, in place of any pre-existing hipoglycaemic therapeutic scheme

SUMMARY:
This work is aimed at improving the quality of life of older patients affected by type 2 diabetes. The investigators will try to amiliorate the complexity of hypogliceamic treatment in a little group of older patients with type 2 diabetes reducing the number of pills and/or insulin administration using a single daily dose of a fixed combination of insulin degludec and liraglutide. This therapeutic semplification will be done indipendently of pre-existent glicaemic control.

DETAILED DESCRIPTION:
Older patients with type 2 diabetes often have numerous coexisting medical problems for which these subjets prescribed multiple medications. Actually, diabetes, hyertension, cardiovascular diseases (CVDs), neurodegenerative diseases (NDDs), digestive and respiratory disorders are common in aged peolple and tend to coexist. Unfortunally, the complex therapy of these diseases increases the risk of adverse drug events. Furthermore, there is marked heterogeneity in health status and functional capacity in older diabetic subjects, often making prescribing decisions complex and challenging. On the other hand, despite of the use of many medicines, undertreatment is also frequent present in the elderly and the probability of underprescription increased significantly with the number of medicines.Both conditions have a detrimental effect on quality of life (QoL) of elderly subjects increasing the risk of disability and death. Therefore, older people should benefit greatly of a simplification of drug regimens and reduction of pill burdens as well as better explanations of the reason for the prescriptions. The combination of insulin degludec (100 units/mL) and liraglutide (3.6 mg/mL), termed IDegLira, was approved in 2014 for the treatment of type 2 diabetes inadequately controlled with oral glucose-lowering agents alone or in combination with a GLP-1 receptor agonist or basal insulin (European indication). Interestingly, RCTs and real-world evidence provided insights into effectiveness and safety in routine clinical practice. However, beyond its known metabolic efficacy IDegLira has a very small hypoglicaemic rate, with a single daily and flexible administration dose and a very good safety profile that makes it suitable for fragile diabetic old patients.

ELIGIBILITY:
Inclusion Criteria:

* frail very old type 2 diabetes patients without severe cognitive impairment and/or grave depression with 3 or more daily hypoglycaemic drug administrations

Exclusion Criteria:

* e-GFR < 15 ml/min
* any experimental clinical trial participation or every experimental drug use in the previous 6 months before commencing this study
* every know or suspected allergic reaction to deglutec or any other GLP-1 agonist
* any known contraindication to IDegLira use (as described in product characteristics)
* Recent cancer diagnosis (<3 y) or active radio- or chemo-therapy. Cancer diagnosis older than 3 years before commencing the study is allowed
* Mini mental state examination score lower than 14/30 and/or Activity Daily Living score lower than 1/6 and/or Instrumenctal Activity Daily Living lower than 1/8

Ages: 75 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Self reported quality of Life (CASP-19) | 6 months
  All participants with treatment-related modification of quality of life as assessed by CASP-19
The Diabetes Treatment Satisfaction (DTSQ) | 6 months
  All participants with treatment-related self reported satisfation for diabetes therapy as assessed by DTSQ

SECONDARY OUTCOMES:
Glycemic control | 6 months
  Glycaemic control evaluated by treatment-related modification of fasting glucose and HbA1c
Hypoglycaemia | 6 months
  Self reported hypoglycaemic events rate
Self reported depression (GDS) | 6 months
  All participants with treatment-related modification of depression as assessed by GDS (Geriatric Depression Scale)
Hypoglycaemic related hospitalizations | 6 months
  Numbers of treatment-related hypoglycaemic hospitalizations
Cognitive function (MMSE) | 6 months
  All participants with treatment-related modification of cognitive function as assessed by Mini Mental State Examination (MMSE)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federici, Professor, Study Chair — Department of Systems Medicine
Locations (1):
- Stefano Rizza, Roma, Italy